CLINICAL TRIAL: NCT00767000
Title: A Phase IIb, Multicenter, Randomized, Double-Blind, Placebo-Controlled Dose-Range Finding Clinical Trial of MK0941 in Patients With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Insulin
Brief Title: Dose Range Finding Study of MK-0941 in Patients With Type 2 Diabetes Mellitus on Insulin (MK-0941-007 AM3 EXT1 AM1)(TERMINATED)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0941-007; 2008_557
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Results first posted 2012-09-03 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-((6-(ethylsulfonyl)-3-pyridinyl)oxy)-5-(2-hydroxy-1-methylethoxy)-N-(1-methyl-1H-pyrazol-3-yl)benzamide; Insulin Glargine; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- MK-0941 10 mg (Experimental)
  Interventions: Drug: MK-0941; Biological: Lantus; Drug: Metformin
- MK-0941 20 mg (Experimental)
  Interventions: Drug: MK-0941; Biological: Lantus; Drug: Metformin
- MK-0941 30 mg (Experimental)
  Interventions: Drug: MK-0941; Biological: Lantus; Drug: Metformin
- MK-0941 40 mg (Experimental)
  Interventions: Drug: MK-0941; Biological: Lantus; Drug: Metformin
- Placebo (Placebo Comparator)
  Interventions: Drug: Comparator: Placebo; Biological: Lantus; Drug: Metformin

INTERVENTIONS:
Drug: MK-0941 — MK-0941 tablets three times daily
  Arms: MK-0941 10 mg; MK-0941 20 mg; MK-0941 30 mg; MK-0941 40 mg
Drug: Comparator: Placebo — Matching placebo to MK-0941 three times daily
  Arms: Placebo
Biological: Lantus — Lantus injection once daily
  Other Names: Insulin glargine injection
Drug: Metformin — Metformin ≥1500 mg/day at a stable dose for at least 6 weeks before Screening and for the duration of the study. The number of randomized participants who receive metformin will be capped at 70% of enrollment.

SUMMARY:
The purpose of this study is to test the effect of MK-0941 as add-on therapy for participants taking insulin for type 2 diabetes mellitus. The primary hypotheses of this study are that treatment with MK-0941 added to insulin will provide greater reduction in hemoglobin A1c (HbA1c) level than will placebo added to insulin at 14 weeks, and that MK-0941 will be well-tolerated at 1 or more doses that demonstrate efficacy.

DETAILED DESCRIPTION:
This study is a 54-week randomized, double-blind base study with an optional 104-week extension study (MK-0941-007-11). Beginning on Week 16, participants not randomized to the maximum dose of MK-0941 could up-titrate to MK-0941 40 mg three times daily. Participants who complete the 54-week base study are eligible to enter the extension study and will remain in the treatment group to which they were assigned in the base study.

ELIGIBILITY:
Inclusion Criteria:

* has type 2 diabetes mellitus
* has body mass index >20 and <43 kg/m^2
* is a male, or a female who is unlikely to conceive
* currently on a stable dose of insulin with or without metformin for Type 2 diabetes mellitus

Extension Study Inclusion Criteria:

* completed the base study either on double-blind study medication or as part of the post-treatment follow up population
* had ≥85% compliance with double-blind and open-label medication during the base study double-blind treatment period

Exclusion Criteria:

* has any history of Type 1 diabetes mellitus or ketoacidosis
* has received more that 1 week of thiazolidinedione (such as pioglitazone or rosiglitazone) therapy or injectable increatin-based therapy (such as Byetta) within the prior 8 weeks
* has had ≥2 episodes during their lifetime or >1 episode within the past year resulting in hypoglycemic seizures, comas, or unconsciousness
* is on a weight loss program and is not in the maintenance phase, or patient is taking a weight loss medication (e.g., orlistat, sibutramine, rimonabant) within 8 weeks of Visit 1
* has undergone surgery within 30 days prior to Visit 1 or has planned major surgery

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 813 (Actual)
Dates: Start 2008-10; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Meininger GE, Scott R, Alba M, Shentu Y, Luo E, Amin H, Davies MJ, Kaufman KD, Goldstein BJ. Effects of MK-0941, a novel glucokinase activator, on glycemic control in insulin-treated patients with type 2 diabetes. Diabetes Care. 2011 Dec;34(12):2560-6. doi: 10.2337/dc11-1200. Epub 2011 Oct 12. PMID 21994424

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-0941 10 mg: MK-0941 10 mg three times daily plus insulin once daily with or without metformin
- MK-0941 20 mg: MK-0941 20 mg three times daily plus insulin once daily with or without metformin
- MK-0941 30 mg: MK-0941 30 mg three times daily plus insulin once daily with or without metformin
- MK-0941 40 mg: MK-0941 40 mg three times daily plus insulin once daily with or without metformin
- Placebo: Placebo three times daily plus insulin once daily with or without metformin
Period: 54-week Study
Arm/Group | MK-0941 10 mg | MK-0941 20 mg | MK-0941 30 mg | MK-0941 40 mg | Placebo
Started | 119 | 117 | 117 | 229 (Includes additional participants enrolled to enhance evaluation of the safety profile of MK-0941) | 231 (Includes additional participants enrolled to enhance evaluation of the safety profile of MK-0941)
Completed | 11 | 4 | 8 | 4 | 7
Not Completed | 108 | 113 | 109 | 225 | 224
Not completed — Adverse Event | 4 | 6 | 6 | 8 | 4
Not completed — Creaninine/creatinine clearance | 2 | 1 | 2 | 2 | 4
Not completed — Hyperglycemia | 0 | 0 | 1 | 0 | 1
Not completed — Hypoglycemia | 0 | 1 | 0 | 0 | 0
Not completed — Interruption of study medication | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 1 | 0 | 5
Not completed — Lost to Follow-up | 4 | 0 | 1 | 4 | 2
Not completed — Physician Decision | 4 | 0 | 1 | 1 | 1
Not completed — Progressive disease | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 5 | 11 | 13
Not completed — Study terminated by sponsor | 90 | 102 | 89 | 196 | 194
Not completed — Reason not reported | 0 | 0 | 0 | 1 | 0
Period: Optional 104-week Extension
Arm/Group | MK-0941 10 mg | MK-0941 20 mg | MK-0941 30 mg | MK-0941 40 mg | Placebo
Started | 7 (The extension study was optional. Not all participants completing the 54-week study continued.) | 3 (The extension study was optional. Not all participants completing the 54-week study continued.) | 7 (The extension study was optional. Not all participants completing the 54-week study continued.) | 2 (The extension study was optional. Not all participants completing the 54-week study continued.) | 4 (The extension study was optional. Not all participants completing the 54-week study continued.)
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 3 | 7 | 2 | 4
Not completed — Study terminated by sponsor | 7 | 3 | 7 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-0941 10 mg | MK-0941 20 mg | MK-0941 30 mg | MK-0941 40 mg | Placebo | Total
Number analyzed (Participants) | 119 | 117 | 117 | 229 | 231 | 813
Age, Customized [Number; unit: participants]
  26 to 71 years | 119 | 117 | 117 | 229 | 231 | 813
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 57 | 54 | 123 | 115 | 416
  Male | 52 | 60 | 63 | 106 | 116 | 397

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1c (HbA1c) Level
Description: Least square means change from baseline in HbA1c. HbA1c represents the percentage of glycated hemoglobin. A negative number means reduction in HbA1c level.
Time Frame: Baseline and Weeks 14, 54, 106, and 158
Population: Full analysis set. The additional participants added to the MK-0941 40 mg and placebo arms to enhance evaluation of safety were not included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent HbA1c
Arm/Group | MK-0941 10 mg | MK-0941 20 mg | MK-0941 30 mg | MK-0941 40 mg | Placebo
Number analyzed (Participants) | 118 | 117 | 117 | 118 | 115
Percent HbA1c
  Week 14 | -0.59 [-0.80 to -0.38] | -0.72 [-0.92 to -0.52] | -0.89 [-1.10 to -0.69] | -0.83 [-1.03 to -0.62] | -0.08 [-0.28 to 0.13]
  Week 54 (no participants analyzed) | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158
  Week 106 (no participants analyzed) | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158
  Week 158 (no participants analyzed) | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158
Statistical Analysis 1: Comparison: MK-0941 10 mg vs Placebo; Analysis for change from baseline to Week 14; Test type: Superiority or Other; p < 0.001, Constrained longitudinal model; Least Squares Mean Difference = -0.51, 95% CI [-0.80 to -0.22]
Statistical Analysis 2: Comparison: MK-0941 20 mg vs Placebo; Analysis for change from baseline to Week 14; Test type: Superiority or Other; p < 0.001, Constrained longitudinal model; Least Squares Mean Difference = -0.64, 95% CI [-0.93 to -0.36]
Statistical Analysis 3: Comparison: MK-0941 30 mg vs Placebo; Analysis for change from baseline to Week 14; Test type: Superiority or Other; p < 0.001, Contrained longitudinal model; Least Squares Mean Difference = -0.81, 95% CI [-1.10 to -0.53]
Statistical Analysis 4: Comparison: MK-0941 40 mg vs Placebo; Analysis for change from baseline to Week 14; Test type: Superiority or Other; p < 0.001, Constrained longitudinal model; Least Squares Mean Difference = -0.75, 95% CI [-1.04 to -0.46]

2. Secondary Outcome: Change in the Two-hour Post Meal Glucose Level
Description: Least squares mean change from baseline in 2-hour post meal glucose level.
Time Frame: Baseline and Weeks 14, 54, 106, and 158
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | MK-0941 10 mg | MK-0941 20 mg | MK-0941 30 mg | MK-0941 40 mg | Placebo
Number analyzed (Participants) | 112 | 114 | 113 | 115 | 111
mg/dL
  Week 14 | -39.0 [-52.0 to -25.1] | -29.2 [-42.5 to -15.9] | -37.4 [-51.2 to -23.6] | -39.3 [-53.1 to -25.5] | -2.4 [-16.0 to 11.2]
  Week 54 (no participants analyzed) | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158
  Week 106 (no participants analyzed) | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158
  Week 158 (no participants analyzed) | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158
Statistical Analysis 1: Comparison: MK-0941 10 mg vs Placebo; Analysis for change from baseline to Week 14; Test type: Superiority or Other; p < 0.001, Constrained longitudial model; Least Squares Mean Difference = -36.6, 95% CI [-55.6 to -17.5]
Statistical Analysis 2: Comparison: MK-0941 20 mg vs Placebo; Analysis for change from baseline to Week 14; Test type: Superiority or Other; p = 0.005, Constrained longitudinal model; Least Squares Mean Difference = -26.7, 95% CI [-45.4 to -8.1]
Statistical Analysis 3: Comparison: MK-0941 30 mg vs Placebo; Analysis for change from baseline to Week 14; Test type: Superiority or Other; p < 0.001, Constrained longitudinal model; Least Squares Mean Difference = -35.0, 95% CI [-54.0 to -16.0]
Statistical Analysis 4: Comparison: MK-0941 40 mg vs Placebo; Analysis for change from baseline to Week 14; Test type: Superiority or Other; p < 0.001, Constrained longitudinal model; Least Squares Mean Difference = -36.9, 95% CI [-55.9 to -17.9]

3. Secondary Outcome: Change in the Fasting Plasma Glucose Level
Description: Least squares mean change from baseline in fasting plasma glucose.
Time Frame: Baseline and Weeks 14, 54, 106, and 158
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | MK-0941 10 mg | MK-0941 20 mg | MK-0941 30 mg | MK-0941 40 mg | Placebo
Number analyzed (Participants) | 118 | 117 | 117 | 118 | 115
mg/dL
  Week 14 | -10.0 [-19.9 to 0.0] | -1.5 [-10.9 to 7.9] | -21.1 [-30.9 to -11.2] | -5.0 [-14.9 to 4.8] | -11.8 [-21.4 to -2.1]
  Week 54 (no participants analyzed) | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158
  Week 106 (no participants analyzed) | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158
  Week 158 (no participants analyzed) | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158 | NA [NA to NA] — Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 54, 106, or 158
Statistical Analysis 1: Comparison: MK-0941 10 mg vs Placebo; Analysis for change from baseline to Week 14; Test type: Superiority or Other; p = 0.791, Constrained longitudinal model; Least Squares Mean Difference = 1.8, 95% CI [-11.6 to 15.2]
Statistical Analysis 2: Comparison: MK-0941 20 mg vs Placebo; Analysis for change from baseline to Week 14; Test type: Superiority or Other; p = 0.121, Constrained longitudinal model; Least Squares Mean Difference = 10.3, 95% CI [-2.7 to 23.2]
Statistical Analysis 3: Comparison: MK-0941 30 mg vs Placebo; Analysis for change from baseline to Week 14; Test type: Superiority or Other; p = 0.169, Constrained longitudinal model; Least Squares Mean Difference = -9.3, 95% CI [-22.6 to 4.0]
Statistical Analysis 4: Comparison: MK-0941 40 mg vs Placebo; Analysis for change from baseline to Week 14; Test type: Superiority or Other; p = 0.321, Constrained longitudinal model; Least Squares Mean Difference = 6.7, 95% CI [-6.6 to 20.0]

4. Secondary Outcome: Percentage of Participants Who Achieve an HbA1c of <7.0%
Time Frame: Weeks 106 and 158
Population: Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 106 or 158
Arm/Group | MK-0941 10 mg | MK-0941 20 mg | MK-0941 30 mg | MK-0941 40 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants Achieving an HbA1c of <7.0% at Week 54 Who Maintain an HbA1c of <7.0%
Time Frame: Weeks 54, 106 and 158
Population: Due to early termination and small numbers of participants, no efficacy analyses were performed at Weeks 106 or 158
Arm/Group | MK-0941 10 mg | MK-0941 20 mg | MK-0941 30 mg | MK-0941 40 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event
Time Frame: Entire study including 54-week study and 104-week extension
Population: Full analysis set. Includes additional participants enrolled in the MK-0941 40 mg and placebo groups to enhance evaluation of the safety profile of MK-0941.
Measure: Number; unit: percentage of participants
Arm/Group | MK-0941 10 mg | MK-0941 20 mg | MK-0941 30 mg | MK-0941 40 mg | Placebo
Number analyzed (Participants) | 119 | 117 | 117 | 229 | 231
percentage of participants | 80.7 | 79.5 | 80.3 | 65.5 | 65.4

7. Primary Outcome: Percentage of Participants Who Discontinued Study Medication Due to an Adverse Event
Time Frame: Entire study including 54-week study and 104-week extension
Measure: Number; unit: percentage of participants
Arm/Group | MK-0941 10 mg | MK-0941 20 mg | MK-0941 30 mg | MK-0941 40 mg | Placebo
Number analyzed (Participants) | 119 | 117 | 117 | 229 | 231
percentage of participants | 3.4 | 5.1 | 6.8 | 3.1 | 1.7

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the entire study including the 54-week study and 104-week extension
Arm/Group | MK-0941 10 mg | MK-0941 20 mg | MK-0941 30 mg | MK-0941 40 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 11/119 | 12/117 | 11/117 | 13/229 | 8/231
Other Adverse Events (participants affected / at risk) | 74/119 | 75/117 | 78/117 | 120/229 | 101/231
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0941 10 mg (N=119) | MK-0941 20 mg (N=117) | MK-0941 30 mg (N=117) | MK-0941 40 mg (N=229) | Placebo (N=231)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cyst rupture (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ovarian mass (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0941 10 mg (N=119) | MK-0941 20 mg (N=117) | MK-0941 30 mg (N=117) | MK-0941 40 mg (N=229) | Placebo (N=231)
Cataract (Eye disorders) | 10 (13) | 12 (16) | 17 (22) | 10 (11) | 20 (20)
Diabetic retinopathy (Eye disorders) | 3 (3) | 6 (8) | 6 (8) | 4 (4) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 7 (9) | 4 (4) | 8 (13) | 11 (22)
Influenza (Infections and infestations) | 6 (7) | 4 (4) | 8 (9) | 10 (14) | 8 (10)
Nasopharyngitis (Infections and infestations) | 8 (10) | 13 (14) | 12 (12) | 12 (16) | 10 (12)
Upper respiratory tract infection (Infections and infestations) | 10 (11) | 6 (7) | 11 (16) | 11 (14) | 6 (7)
Hypoglycaemia (Metabolism and nutrition disorders) | 57 (425) | 58 (475) | 57 (719) | 94 (690) | 67 (350)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1) | 1 (1) | 3 (3) | 6 (6)
Headache (Nervous system disorders) | 4 (8) | 12 (12) | 5 (6) | 13 (16) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.